CLINICAL TRIAL: NCT00871897
Title: Cognitive Benefits of Cardiac Rehabilitation in Heart Failure
Brief Title: Examining the Cognitive Benefits of Cardiac Rehabilitation in People With Heart Failure (The CHF CaRe Study)
Acronym: CHF CaRe
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: John Gunstad, PhD, Assistant Professor, Kent State University
Other Study IDs: 649; R01HL089311 (NIH)
Record Dates: First submitted 2009-03-27; First posted 2009-03-30 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2009-12

CONDITIONS: Heart Failure
Keywords: Neuropsychology; Cardiac Rehabilitation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cardiac Rehabilitation: People with heart failure who elect to participate in cardiac rehabilitation.
- No Cardiac Rehabiliation: People with heart failure who elect NOT to participate in cardiac rehabilitation.

SUMMARY:
People with heart failure may experience problems with cognitive function, including memory and attention. Cardiac rehabilitation, which is an individualized program for heart failure patients that aims to improve their heart health, may also improve cognitive function. This study will examine the relationship between heart failure and cognitive function and how undergoing cardiac rehabilitation affects cognitive function in older adults with heart failure.

DETAILED DESCRIPTION:
Over 5 million people in the United States have heart failure, and 500,000 more develop this condition each year. Up to 80% of people with heart failure experience cognitive functioning difficulties, including problems with memory, attention, and other thinking skills. People with heart failure often participate in a cardiac rehabilitation program, which is an individualized program that aims to improve a person's physical and mental health while dealing with a heart-related condition. Cardiac rehabilitation is different for each person, but it can include medical counseling on how to manage a heart condition and how to modify risk factors for further heart problems, including lowering blood pressure and cholesterol levels, stopping smoking, and losing weight. Nutritional counseling and an exercise program may also be a part of cardiac rehabilitation. Preliminary research has shown that people with heart failure who participate in a cardiac rehabilitation program may experience improved cognitive function. This is thought to be a result of increased blood flow to the brain and improved autonomic nervous system function, which is responsible for regulating various body functions. In this study, researchers will explore the relationship between heart failure and cognitive function, examine how cognitive function changes over time in heart failure patients, and evaluate how cardiac rehabilitation may affect cognitive function in older adults. Specifically, researchers will examine how physical activity and patterns of blood flow affect cognitive function.

This study will enroll people with heart failure who are participating in a 12-week cardiac rehabilitation program and people with heart failure who are not participating in a cardiac rehabilitation program. All participants will attend study visits at baseline, Week 12, and Month 12. At each study visit, participants will undergo neuropsychological testing, heart rate and blood pressure measurements, and a walking exercise test. They will also complete questionnaires to assess diet, physical activity, and stress levels. Participants will undergo an imaging procedure to measure blood flow in the neck and head, and some participants will also undergo a magnetic resonance imaging (MRI) procedure of their brain. For 1 week after each study visit, participants will wear a physical activity monitor. At Months 6 and 9, participants will complete questionnaires and mail these back to study researchers.

The study completion date listed in this record was obtained from the "Completed Date" entered in the Query View Report System (QVR).

ELIGIBILITY:
Inclusion Criteria:

* Systolic heart failure confirmed by perfusion stress scan

Exclusion Criteria:

* Has a pacemaker

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with heart failure
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-04; Primary Completion 2012-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Gunstad, PhD, Principal Investigator — Kent State University
Locations (1):
- Summa Health System, Akron, Ohio, United States

REFERENCES:
- [Derived] Walter FA, Gathright E, Redle JD, Gunstad J, Hughes JW. Depressive Symptoms are Associated with Heart Rate Variability Independently of Fitness: A Cross-Sectional Study of Patients with Heart Failure. Ann Behav Med. 2019 Oct 7;53(11):955-963. doi: 10.1093/abm/kaz006. PMID 30958884
- [Derived] Alosco ML, Spitznagel MB, van Dulmen M, Raz N, Cohen R, Sweet LH, Colbert LH, Josephson R, Hughes J, Rosneck J, Gunstad J. Cognitive function and treatment adherence in older adults with heart failure. Psychosom Med. 2012 Nov-Dec;74(9):965-73. doi: 10.1097/PSY.0b013e318272ef2a. Epub 2012 Oct 31. PMID 23115344